CLINICAL TRIAL: NCT04506463
Title: A Phase IIb, Randomized, Double-Blind, Placebo-Controlled, Single-administration, Multiple-Dose Study to Demonstrate the Efficacy and Safety of MM-II for Treatment of Knee Pain in Subjects With Symptomatic Knee Osteoarthritis
Brief Title: Efficacy and Safety of MM-II for Treatment of Knee Pain in Subjects With Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Collaborators: Moebius Medical Ltd. (Industry); Nordic Bioscience Clinical Development (NBCD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_17_17
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-06

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental): MM-II 1 ml
  Interventions: Drug: MM-II dose I
- Arm B (Experimental): MM-II 3 ml
  Interventions: Drug: MM-II dose II
- Arm C (Experimental): MM-II 6 ml
  Interventions: Drug: MM-II dose III
- Arm 4 (Placebo Comparator): Placebo 1ml
  Interventions: Drug: Placebo
- Arm 5 (Placebo Comparator): Placebo 3ml
  Interventions: Drug: Placebo
- Arm 6 (Placebo Comparator): Placebo 6ml
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MM-II dose I — Intra-articular injection
  Arms: Arm A
Drug: MM-II dose II — Intra-articular injection
  Arms: Arm B
Drug: MM-II dose III — Intra-articular injection
  Arms: Arm C
Drug: Placebo — Intra-articular injection
  Arms: Arm 4
Drug: Placebo — Intra-articular injection
  Arms: Arm 5
Drug: Placebo — Intra-articular injection
  Arms: Arm 6

SUMMARY:
This is a phase IIb, randomized, double-blind, placebo-controlled study to determine the efficacy and safety of MM-II in subjects with symptomatic knee OA as compared to matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to provide written consent, understand study requirements, is prepared to complete study procedures and is able to independently communicate meaningfully with study personnel
2. Presence of index knee pain for at least 6 months prior to Screening
3. Men or women ≥ 40 years of age at the time of Screening
4. Radiographic evidence of knee Osteoarthritis

Exclusion Criteria:

1. Pain in the contralateral knee with a severity of ≥ 30 mm on a 100 mm VAS
2. Presence of ≥ 40 mm on a 100 mm VAS pain in any other joints
3. Concomitant moderate or large size synovial fluid effusion of the index knee at Screening .
4. Known diagnosis of infection in the index knee in the past five years prior to Screening

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (21):
  - Sunpharma site no. 20, Birmingham, Alabama
  - Sunpharma site no. 11, Tempe, Arizona
  - Sunpharma site no. 25, Riverside, California
  - Sunpharma site no. 26, San Diego, California
  - Sunpharma site no. 06, Stamford, Connecticut
  - Sunpharma site no. 10, Lady Lake, Florida
  - Sunpharma site no. 08, Lake Worth, Florida
  - Sunpharma site no. 13, Maitland, Florida
  - Sunpharma site no. 22, Miami, Florida
  - Sunpharma Site no 27, Miami, Florida
  - Sunpharma site no. 12, Miami, Florida
  - SunPharma Site no 23, Miami, Florida
  - Sunpharma site no. 05, Sunrise, Florida
  - Sunpharma site no. 04, The Villages, Florida
  - Sunpharma site no. 18, Flossmoor, Illinois
  - Sunpharma site no. 07, Hazelwood, Missouri
  - Sunpharma site no. 17, Williamsville, New York
  - Sunpharma site no. 19, Edmond, Oklahoma
  - Sunpharma site no. 09, Charleston, South Carolina
  - SunPharma Site No 24, Columbia, South Carolina
  - Sunpharma site no. 21, Fort Mill, South Carolina
- Denmark (3):
  - Sunpharma site no. 02, Gandrup
  - Sunpharma site no. 01, Herlev
  - Sunpharma site no. 03, Vejle
- Sunpharma site no. 14, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: MM-II 1 ml: MM-II 1 ml
  MM-II dose I: Intra-articular injection
- Arm B: MM-II 3 ml: MM-II 3 ml
  MM-II dose II: Intra-articular injection
- Arm C: MM-II 6 ml: MM-II 6 ml
  MM-II dose III: Intra-articular injection
- Arm 4: Placebo 1 ml: Placebo 1 ml
  Placebo: Intra-articular injection
- Arm 5: Placebo 3 ml: Placebo 3 ml
  Placebo: Intra-articular injection
- Arm 6: Placebo 6 ml: Placebo 6 ml
  Placebo: Intra-articular injection
Period: Overall Study
Arm/Group | Arm A: MM-II 1 ml | Arm B: MM-II 3 ml | Arm C: MM-II 6 ml | Arm 4: Placebo 1 ml | Arm 5: Placebo 3 ml | Arm 6: Placebo 6 ml
Started | 103 | 83 | 76 | 28 | 79 | 28
Completed | 98 | 80 | 66 | 27 | 71 | 27
Not Completed | 5 | 3 | 10 | 1 | 8 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 4: Placebo 1ml: Placebo 1ml
  Placebo: Intra-articular injection
- Arm 5: Placebo 3ml: Placebo 3ml
  Placebo: Intra-articular injection
- Arm 6: Placebo 6ml: Placebo 6ml
  Placebo: Intra-articular injection
- Total: Total of all reporting groups
Arm/Group | Arm A: MM-II 1 ml | Arm B: MM-II 3 ml | Arm C: MM-II 6 ml | Arm 4: Placebo 1ml | Arm 5: Placebo 3ml | Arm 6: Placebo 6ml | Total
Number analyzed (Participants) | 103 | 83 | 76 | 28 | 79 | 28 | 397
Age, Customized [Number; unit: participants]
  ≤ 65 Years | 65 | 41 | 52 | 19 | 50 | 15 | 242
  > 65 Years | 38 | 42 | 24 | 9 | 29 | 13 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 58 | 39 | 20 | 51 | 19 | 258
  Male | 32 | 25 | 37 | 8 | 28 | 9 | 139
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 16 | 3 | 8 | 5 | 59
  Not Hispanic or Latino | 89 | 70 | 60 | 25 | 71 | 23 | 338
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 29 | 19 | 17 | 5 | 21 | 5 | 96
  United States | 27 | 37 | 32 | 10 | 27 | 14 | 147
  Denmark | 47 | 27 | 27 | 13 | 31 | 9 | 154

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A Pain Score
Description: The pain score is based on a score of 0 to 4; the higher the score, the higher the amount of pain.
Time Frame: Week 12
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Arm 6: Placebo 6 ml: Placebo 6ml
  Placebo: Intra-articular injection
Arm/Group | Arm A: MM-II 1 ml | Arm B: MM-II 3 ml | Arm C: MM-II 6 ml | Arm 4: Placebo 1 ml | Arm 5: Placebo 3 ml | Arm 6: Placebo 6 ml
Number analyzed (Participants) | 103 | 83 | 76 | 28 | 78 | 28
score on a scale | -1.28 (0.079) | -1.35 (0.086) | -1.14 (0.092) | -0.96 (0.143) | -1.11 (0.089) | -1.10 (0.142)
Statistical Analysis 1: Comparison: Arm A: MM-II 1 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.850, Mixed Models Analysis
Statistical Analysis 2: Comparison: Arm B: MM-II 3 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.085, Mixed Models Analysis
Statistical Analysis 3: Comparison: Arm C: MM-II 6 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.850, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in Weekly Average of Daily Knee Pain Scores by VAS
Description: Knee pain will be assessed on a score of 0 to 100; the lower on the scale, the less the amount of knee pain experienced. Weekly post-baseline average daily knee pain scores will be calculated.
Time Frame: Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Arm 4: Placebo 1 ml: Placebo 1ml
  Placebo: Intra-articular injection
- Arm 5: Placebo 3 ml: Placebo 3ml
  Placebo: Intra-articular injection
Arm/Group | Arm A: MM-II 1 ml | Arm B: MM-II 3 ml | Arm C: MM-II 6 ml | Arm 4: Placebo 1 ml | Arm 5: Placebo 3 ml | Arm 6: Placebo 6 ml
Number analyzed (Participants) | 103 | 83 | 76 | 28 | 78 | 28
score on a scale | -30.4 (2.81) | -34.5 (3.08) | -23.1 (3.26) | -28.2 (5.19) | -22.7 (3.20) | -30.0 (5.15)
Statistical Analysis 1: Comparison: Arm A: MM-II 1 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.062, Mixed Models Analysis
Statistical Analysis 2: Comparison: Arm B: MM-II 3 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.007, Mixed Models Analysis
Statistical Analysis 3: Comparison: Arm C: MM-II 6 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.936, Mixed Models Analysis

3. Secondary Outcome: Change From Baseline in Weekly Average of Daily Global Pain Scores by VAS
Description: Global pain will be assessed on a score of 0 to 100; the lower on the scale, the less the amount of global pain experienced. Weekly post-baseline average daily global pain scores will be calculated
Time Frame: Week 26
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm A: MM-II 1 ml | Arm B: MM-II 3 ml | Arm C: MM-II 6 ml | Arm 4: Placebo 1 ml | Arm 5: Placebo 3 ml | Arm 6: Placebo 6 ml
Number analyzed (Participants) | 103 | 83 | 76 | 28 | 78 | 28
score on a scale | -21.0 (3.12) | -22.1 (3.54) | -14.4 (3.69) | -17.6 (5.86) | -12.2 (3.55) | -26.3 (6.15)
Statistical Analysis 1: Comparison: Arm A: MM-II 1 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.042, Mixed Models Analysis
Statistical Analysis 2: Comparison: Arm B: MM-II 3 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.037, Mixed Models Analysis
Statistical Analysis 3: Comparison: Arm C: MM-II 6 ml vs Arm 5: Placebo 3 ml; Test type: Superiority; p = 0.648, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 27 week
Description: Safety was assessed using the Safety Analysis Set.The Safety Analysis Set will include all randomized subjects who received the single dose of IP.
  Note:Two subjects were randomized to 6 mL MM-II but received 3 mL MM-II; One subject was randomized to 1 mL MM-II but received 3 mL MM-II
Arm/Group | Arm A: MM-II 1 ml | Arm B: MM-II 3 ml | Arm C: MM-II 6 ml | Arm 4: Placebo 1 ml | Arm 5: Placebo 3 ml | Arm 6: Placebo 6 ml
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/86 | 0/74 | 0/28 | 0/78 | 0/28
Serious Adverse Events (participants affected / at risk) | 4/102 | 0/86 | 3/74 | 0/28 | 3/78 | 1/28
Other Adverse Events (participants affected / at risk) | 75/102 | 49/86 | 49/74 | 15/28 | 46/78 | 19/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: MM-II 1 ml (N=102) | Arm B: MM-II 3 ml (N=86) | Arm C: MM-II 6 ml (N=74) | Arm 4: Placebo 1 ml (N=28) | Arm 5: Placebo 3 ml (N=78) | Arm 6: Placebo 6 ml (N=28)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Esophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 | 0 | 0 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Blood loss anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 (2) | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: MM-II 1 ml (N=102) | Arm B: MM-II 3 ml (N=86) | Arm C: MM-II 6 ml (N=74) | Arm 4: Placebo 1 ml (N=28) | Arm 5: Placebo 3 ml (N=78) | Arm 6: Placebo 6 ml (N=28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5) | 10 (12) | 1 (1) | 6 (8) | 3 (3)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 | 4 (4) | 1 (1)
Injection site joint pain (General disorders) | 0 | 2 (2) | 2 (2) | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
COVID-19 (Infections and infestations) | 18 (18) | 7 (7) | 7 (7) | 4 (4) | 8 (8) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (8) | 3 (3) | 6 (6) | 1 (1) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Root canal infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 3 (3) | 0 | 2 (2) | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 | 3 (3) | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 1 (1) | 1 (1) | 2 (2) | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mandibular mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 1 (2) | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 2 (2) | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 (0) | 0
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 6 (6) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 3 (3) | 2 (2) | 0 | 4 (4) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 | 2 (2) | 0 | 3 (3) | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 4 (4) | 3 (3) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 3 (4) | 0 | 0 | 0 | 1 (1) | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 1 (1) | 0 | 0 | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0
Cataract operation complication (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Buttock injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 (2) | 1 (2) | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 (2) | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0
Influenza like illness (General disorders) | 5 (6) | 1 (1) | 2 (2) | 3 (3) | 3 (4) | 1 (1)
Chest pain (General disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Pyrexia (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
White blood cells urine (Investigations) | 3 (3) | 0 | 0 | 0 | 1 (1) | 0
Hepatic enzyme increased (Investigations) | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 2 (2) | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Electrocardiogram QT interval normal (Investigations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Platelet count increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (2)
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Gamma-glutamyltran sferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 (1) | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (11) | 4 (4) | 2 (2) | 8 (8) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 | 1 (1) | 0
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 (3) | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 0 | 1 (1) | 0 | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 | 2 (2) | 0 | 4 (4) | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 | 1 (1) | 0 | 0 | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 | 1 (1) | 2 (2) | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Hypertension (Vascular disorders) | 8 (8) | 3 | 3 | 0 | 3 (4) | 0
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Age-related macular degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalassaemia minor (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT04506463/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT04506463/SAP_001.pdf